CLINICAL TRIAL: NCT02194842
Title: A Randomized Multicenter Phase III Trial Comparing Enzalutamide vs. a Combination of Ra223 and Enzalutamide in Asymptomatic or Mildly Symptomatic Castration Resistant Prostate Cancer Patients Metastatic to Bone.
Brief Title: Phase III Radium 223 mCRPC-PEACE III
Acronym: PEACE III
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Bayer (Industry); Astellas Pharma Europe Ltd. (Industry); UNICANCER (Other); Canadian Urologic Oncology Group (Other); Latin American Cooperative Oncology Group (Other); Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1333-GUCG; 2014-001787-36 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: metastatic; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Radium-223; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzalutamide (Active Comparator): Enzalutamide will be given at a dose of 160 mg daily
  Interventions: Drug: Enzalutamide
- Enzalutamide and Ra223 (Experimental): Ra223 will be administered 55kBq/kg standard dose monthly for 6 months and given in combination with enzalutamide at a dose of 160 mg daily.
  Interventions: Drug: Ra223; Drug: Enzalutamide

INTERVENTIONS:
Drug: Ra223
  Arms: Enzalutamide and Ra223
Drug: Enzalutamide

SUMMARY:
The primary objective of the trial is to assess if upfront combination of enzalutamide and Ra223 improves radiological progression-free survival (rPFS1) by investigator assessment compared to enzalutamide single agent in castration resistant prostate cancer (CRPC) patients metastatic to bone

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma
* Asymptomatic or mildly symptomatic (defined as short form question #3 in Brief Pain Inventory worst pain must be < 4, see Appendix E)
* Metastatic to bone with ≥ 4 bone metastases (ambiguous areas of increased uptake on 99mTc Bone Scan (BS) should be confirmed by CT or MRI) with or without additional lymph node metastases.

Patients with visceral metastases are not allowed. Patients with multifocal bone lesions are allowed; while patients with diffuse confluent bone lesions (superscan) are not allowed in the trial.

* Note: Patients must start treatment with a bone protecting agent (at doses used to reduce the incidence of skeletal related events) ideally before or at the time of randomization, if patient is not already on one. A minimum of two doses is recommended before the first administration of Ra223 in the experimental arm. The first administration of Ra223 should be scheduled at least 6 weeks after the first administration of bone protecting agent.
* Note: For French sites only, patients must not have undergone a PET/CT scan for restaging prostate cancer using radiopharmaceuticals such as 18F-FDG, 18F-fluoride, 18F-Fluorocholine or a PSMA (prostate-specific membrane antigen) ligand or any other tracer.
* Progressive CRPC according to Prostate Cancer Working Group 3 (PCWG3) (Ref. 22) i.e. either:
* For patients who manifest disease progression solely as a rising PSA level, PCWG3 criteria require documentation of a sequence of rising PSA values at a minimum of 1-week intervals with the last value > 2 ng/mL
* For patients with disease progression manifest in the bone, irrespective of progression by rising PSA, PCWG3 guidelines require appearance of 2 or more new lesions. Ambiguous results should be confirmed by other imaging modalities than bone scan (e.g.: CT-scan or MRI)
* For patients with disease progression manifest at nodal sites, irrespective of progression by rising PSA, PCWG3 requires progression according to RECIST 1.1
* Ongoing androgen deprivation therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonist or antagonist or bilateral orchiectomy
* No known central nervous system metastases or leptomeningeal tumor spread.
* Patients must be at least 18 years old
* WHO Performance status 0-1(see Appendix C)
* Charlson score ≤ 3 (see Appendix G)
* T-score ≥ -2.5 on a DXA scan done in the past 12 months Note: For French sites only, DXA scan done within 6 weeks of randomization
* Castrate serum levels of testosterone < 50 ng/dL
* Biochemistry and hematology:
* Adequate bone marrow function (absolute neutrophil count (ANC) ≥ 1.5 109/L; platelets ≥100 109/L, and hemoglobin ≥ 10.0 g/dL)
* Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN), except for patient with Gilbert's disease where ≤ 5.0 × ULN applies
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN
* Albumin > 25 g/L
* Normal cardiac function according to local standard by 12-lead ECG (complete, standardized 12-lead recording)
* No significant cardiovascular disease including:
* Myocardial infarction within 6 months prior to screening
* Uncontrolled angina within 3 months prior to screening
* Congestive heart failure New York Heart Association (NYHA) class III or IV, or patients with history of congestive heart failure NYHA class III or IV in the past, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%
* History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
* History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
* Uncontrolled hypertension as indicated by a resting systolic blood pressure > 140 millimeters of mercury (mm Hg) or diastolic blood pressure > 90 mm Hg at screening.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to randomization. Blood pressure must be re-assessed on two occasions that are separated by a minimum of 1 hour. The mean SBP / DBP values from all blood pressure assessment timepoints must be ≤140/90 mm Hg in order for a patient to be eligible for the study.

* Hypotension as indicated by systolic blood pressure < 86 mm Hg at screening
* Bradycardia as indicated by a heart rate of < 45 beats per minute on the screening ECG and on physical examination
* Uncontrolled hyperglycemia as indicated by a fasting glucose ≥ 7 mmol/L
* Able to swallow the study drug and comply with study requirements
* Prior or concomitant therapy
* Prior docetaxel is permitted if given in the castration sensitive state and if it was started within 4 months of ADT initiation Note: patients having received docetaxel for CRPC are excluded.
* Prior use of abiraterone is permitted if the patient had a response or stable disease on abiraterone for a minimum of 1 year for metastatic castration sensitive prostate cancer
* Note: patients having received abiraterone for CRPC are excluded. Prior treatment with abiraterone is allowed if it was stopped at least 4 weeks prior to randomization
* No prior treatment with enzalutamide, apalutamide, darolutamide or Ra223
* No concomitant treatment with Cyp17 inhibitors (abiraterone, orteronel) and ketoconazole
* Previous treatment with bicalutamide or flutamide is allowed if it was stopped at least 48 hours prior to randomization
* Corticosteroids are allowed only at a dose ≤ 10 mg of prednisone (or equivalent) no matter the indication
* No prior hemibody external radiotherapy. Patients who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count and platelets
* No prior therapy with other radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188)
* No involvement in another therapeutic trial involving an experimental drug
* No anticancer therapy (except ADT) or treatment with another investigational agent within the last 4 weeks prior to randomization
* No known hypersensitivity to compounds related to enzalutamide or Ra223 (refer to Investigator's brochures)
* No prior history of malignancies other than prostate adenocarcinoma (except patients with basal cell, squamous cell carcinoma of the skin, in-situ carcinoma or low-grade superficial bladder cancer), or the patient has been free of malignancy for a period of 3 years prior to randomization date
* No history of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attack within 12 months of randomization, OR any condition that may pre-dispose to seizure (e.g., prior stroke, brain arterio-venous malformation, head trauma with loss of consciousness requiring hospitalization)
* Drugs known to lower the seizure threshold or prolong QT interval are not permitted (refer to section 5.9.3.2)
* No major surgery within 4 weeks prior to treatment
* No drug or alcohol abuse
* No other serious illness or medical condition, such as but not limited to:
* Any infection ≥ Grade 2 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4
* No gastrointestinal disorder affecting absorption (e.g., gastrectomy or active peptic ulcer disease)
* Crohn's disease or ulcerative colitis
* Osteonecrosis of the jaw
* Any bone disease with an osteoblastic activity
* Bone marrow dysplasia
* Fecal incontinence
* Life-threatening illness unrelated to cancer
* No condition which, in the investigator's opinion, makes the patient unsuitable for trial participation
* Participants who have pregnant partners must use a condom and those with partners of childbearing potential must use a condom and another adequate birth control measure if engaging in sexual activities during the study treatment period and for at least 3 months after last dose of enzalutamide and 6 months after the last dose of Ra223. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations
* For participation in translational research, specific consent must be given. Important note: All eligibility criteria must be adhered to, in case of deviation discussion with EORTC Headquarters and study coordinator is mandatory

Exclusion Criteria:

* No known history of central nervous system metastases or leptomeningeal tumor spread.
* No significant cardiovascular disease including:

  1. Myocardial infarction within 6 months prior to screening
  2. Uncontrolled angina within 3 months prior to screening
  3. Congestive heart failure New York Heart Association (NYHA) class III or IV, or patients with history of congestive heart failure NYHA class III or IV in the past, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%
  4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  5. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  6. Uncontrolled hypertension as indicated by a resting systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening
  7. Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mm Hg) at screening
  8. Bradycardia as indicated by a heart rate of < 45 beats per minute on the screening ECG and on physical examination
* patients having received docetaxel for CRPC are excluded.
* No prior treatment with enzalutamide or Ra223
* No prior and concomitant treatment with Cyp17 inhibitors (abiraterone, orteronel) and ketoconazole
* No prior hemibody external radiotherapy. Patients who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for hemoglobin, absolute neutrophil count and platelets
* No prior therapy with other radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188)
* No involvement in another therapeutic trial involving an experimental drug
* No anticancer therapy or treatment with another investigational agent within the last 4 weeks prior to randomization
* No known hypersensitivity to compounds related to enzalutamide or Ra223
* No prior history of malignancies other than prostate adenocarcinoma (except patients with basal cell, squamous cell carcinoma of the skin, in-situ carcinoma or low-grade superficial bladder cancer), or the patient has been free of malignancy for a period of 3 years prior to randomization date
* No history of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attack within 12 months of enrollment (registration date), or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arterio-venous malformation, head trauma with loss of consciousness requiring hospitalization)
* No major surgery within 4 weeks prior to treatment
* No intake of narcotic analgesia for bone pain
* No drug or alcohol abuse
* No other serious illness or medical condition, such as but not limited to:

  1. Any infection ≥ Grade 2 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4
  2. No gastrointestinal disorder affecting absorption (e.g., gastrectomy or active peptic ulcer disease)
  3. Crohn's disease or ulcerative colitis
  4. Bone marrow dysplasia
  5. Fecal incontinence
  6. Life-threatening illness unrelated to cancer
* No condition which, in the investigator's opinion, makes the patient unsuitable for trial participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
radiological progression-free survival | 46 months after first patient entry
  Radiological progression free survival (rPFS1) is defined according to the recommendations of the "Prostate-Cancer clinical trials Working Group" version 3 and referred to as the "PCWG3"; for the setting "delay/prevent" progression.
  An event of progression according to their definition is either of:
  * Objective progression of the disease according to RECIST 1.1 criteria for soft tissue lesions
  * A skeletal radiological progression defined as the appearance of ≥ 2 new bone lesions and for the first follow-up assessment only (i.e., within 12 weeks ± 1 week, during the flare period), a confirmatory scan performed ≥ 6 weeks later that shows a minimum of two or more additional new lesions (2+2 criterion) In this protocol: PSA progression is not considered disease progression and should NOT trigger a change of treatment.
  The rPFS1 endpoint is subject to a retrospective Blinded Independent Central Review
progression-free survival per Blinded Independent Central Review (PFS1B) | 96 months after first patient entry
  PFS1 per BICR will be defined and analyzed in the same manner as the primary endpoint rPFS1 by investigator assessment. The central reviewers will provide timepoint assessments of skeletal and nonskeletal progression and determinations of respective progression dates from which PFS1 per BICR will be calculated.

SECONDARY OUTCOMES:
Overall survival | 63 months after first patient entry
  number of participants
prostate cancer specific survival | 63 months after first patient entry
  number of participants
Time to First symptomatic skeletal event (TTSSE) | 46 and 63 months after first patient entry
  number of participants
Time to first skeletal progression | 46 and 63 months after first patient entry
  number of months
Time from entry to initiation of next systemic anti-neoplastic therapy (TTNT) | 46 and 63 months after first patient entry
  number of participants
Progression-free survival on second line of treatment (PFS2) | 46 and 63 months after first patient entry
  number of participants
Patient self-rate scale assessing the pain associated to prostate cancer | 46 and 63 months after first patient entry
  Brief Pain Inventory questionnaire: BPI questionnaire is a validated instrument that is a patient self-rated scale assessing level of pain, effect of the pain on activities of daily living, and analgesic use. The BPI also measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. The short form of the BPI is used in this study. It is intended to capture two dimensions of pain: severity and interference. This short version of the BPI contains four pain severity items and seven pain interference items rated on 0-10 scales and uses a 24-hour recall period.
Time to pain progression (TTPP) | 63 months after first patient entry
  defined as an increase of 2 or more points in the "worst pain in 24 hours" score from baseline observed at 2 consecutive evaluations ≥ 4 weeks apart OR initiation of short or long-acting opioid use for pain
Occurence of adverse events | 63 months after first patient entry
  Adverse events will be graded according to the "Common Terminology Criteria for Adverse events" CTCAE, version 4.0
Time to opiate use for cancer-related pain | 63 months after first patient entry
  number of participants
Patient self-rate scale assessing the Quality of Life | 46 and 63 months after first patient entry
  EQ5D-5L questionnaire asks respondents to simply 'mark an X on the scale to indicate how your health is TODAY' and then to 'write the number you marked on the scale in the box below'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
  The respondent is asked to indicate his health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. It should be noted that the numerals 1-5 have no arithmetic properties and should not be used as a cardinal score.
rate of skeletal fractures | 63 months after first patient entry
  The rate of skeletal fractures per patient/year of follow-up will be estimated in each treatment arm using recurrent-event analysis methods. Analyses by type of fracture (e.g. pathological fracture) will also be conducted as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Tombal, Prof, Study Chair — Cliniques Universitaires de Saint Luc; Silke Gillessen, Prof, Study Chair — Oncology Institute of Southern Switzerland - Ospedale San Giovanni
Locations (64):
- Belgium (8):
  - Hopital Universitaire Brugmann, Brussels
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Groeninge Kortrijk, Kortrijk
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - AZ Turnhout, Turnhout
  - CHU Dinant Godinne - UCL Namur, Yvoir
- Brazil (13):
  - Hospital de Amor, Barretos
  - Hospital Erasto Gaertner, Curitiba
  - Centro Pesquisas Oncologicas, Florianópolis
  - Oncocentro, Fortaleza
  - Hospital Moinhos de Vento, Porto Alegre
  - Centro de Pesquisas Clinicas em Oncologia - Hospital Sao Lucas, Porto Alegre
  - Instituto de Medicina Integral Professor Fernando Figueira - IMIP, Recife
  - Centro de Tratamentos de Tumores Botafogo, Rio de Janeiro
  - Clínica Oncológica - CLION, Salvador
  - Centro de Estudos e Pesquisa Hematologia e Oncologia, Santo André
  - Hospital Beneficencia Portuguesa, São Paulo
  - Hospital Paulistano, São Paulo
  - Sao Camilo Oncologia - Instituto Brasileiro de Controle do Cancer, São Paulo
- Canada (8):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Hamilton And District Urology Association, Hamilton, Ontario
  - London Regional Cancer Center, London, Ontario
  - Odette Cancer Centre - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Oci Princess Margaret Hospital, Toronto, Ontario
  - Centre de sante et de services sociaux de Chicoutimi, Chicoutimi, Quebec
  - CHUM - Centre Hospitalier de l'Université de Montreal - Pavillon Saint-Luc, Montreal, Quebec
  - Chuq-Pavillon Hotel-Dieu De Quebec, Québec, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Paul Papin, Angers
  - Centre Francois Baclesse, Caen
  - Assistance Publique - Hopitaux de Paris - CHU Henri Mondor, Créteil
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Saint-Herblain
  - Hopitaux Universitaires de Strasbourg - Hôpitaux Universitaires de Strasbourg - Hôpital civil, Strasbourg
  - Gustave Roussy, Villejuif
- Ireland (3):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - Tallaght University Hospital, Dublin
- Italy (3):
  - Ospedale B.Ramazzini, Carpi
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
- Norway (2):
  - Soerlandet Sykehus-Kristiansand, Kristiansand
  - University Hospital of North Norway, Tromsø
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Spain (10):
  - Hospital Del Mar, Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario QuironSalud, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
- Switzerland (3):
  - Oncology Institute of Southern Switzerland - Ospedale San Giovanni, Bellinzona
  - Kantonsspital St Gallen, Sankt Gallen
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (4):
  - United Lincolnshire Hospitals NHS Trust - Lincoln County Hospital, Lincoln
  - Royal Marsden Hospital - Chelsea, London, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham

REFERENCES:
- [Derived] Tombal B, Saad F, Gallardo E, Soares A, Loriot Y, McDermott R, Briers E, Lagstrom M, Coens C, Poncet C, Fournier B, Gillessen S. A plain language summary of the EORTC 1333/PEACE-3 study of enzalutamide alone vs enzalutamide plus radium-223 in patients with metastatic castrationresistant prostate cancer (mCRPC) and bone metastases. Future Oncol. 2025 Dec;21(30):3845-3858. doi: 10.1080/14796694.2025.2592722. Epub 2025 Nov 28. PMID 41313045
- [Derived] Gillessen S, Tombal B, Turco F, Choudhury A, Rodriguez-Vida A, Gallardo E, Velho PI, Nole F, Cruz F, Loriot Y, McDermott R, Roumeguere T, Daugaard G, Yamamura R, Bompas E, Maroto P, Polo MH, da Trindade KM, Preto DD, Skoneczna I, Lecouvet F, Coens C, Fournier B, Saad F. Decrease in Fracture Rate with Mandatory Bone-protecting Agents in the EORTC 1333/PEACE-3 Trial Comparing Radium-223 Combined with Enzalutamide Versus Enzalutamide Alone: A Safety Analysis. Eur Urol. 2025 Mar;87(3):285-288. doi: 10.1016/j.eururo.2024.11.027. Epub 2025 Jan 17. PMID 39827019